CLINICAL TRIAL: NCT06940882
Title: Development and Exploration of the Acceptability and Feasibility of a Novel Screening Tool for Anosognosia After Stroke, Designed for Routine Use in Hospital Settings.
Brief Title: Development of a Novel Screening Tool for Anosognosia After Stroke.
Status: Not yet recruiting | Type: Observational
Sponsor: University of Exeter (Other)
Collaborators: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 24-25-17
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Anosognosia; Stroke
Keywords: Anosognosia; Stroke; Assessment
MeSH Terms: conditions — Agnosia; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients admitted to a stroke rehabilitation unit following clinical diagnosis of stroke. Participation will involve completion of a new screening tool for anosognosia, to be administered by multi-disciplinary staff working on the stroke rehabilitation unit.
- Staff: Multi-disciplinary staff working on a stroke rehabilitation unit. Participation will involve administering a new screening tool for anosognosia with patients, and then attending focus groups to explore the acceptability and feasibility of the new screening tool among the staff group.

SUMMARY:
Anosognosia, a neurological inability to acknowledge or comprehend one's own (dis)abilities, is a multi-faceted phenomenon which has consistently gained traction in research fields spanning psychology, neurology, and cognition since its conceptual introduction in 1914. Though anosognosia is not limited to following only neurological disease or injury, the majority of research has focused on the prevalence and mechanisms of anosognosia after stroke. Despite this, there is no clear consensus among the literature, and thus in clinical practice, as to how anosognosia after stroke should be assessed. This is startling given the plethora of studies which highlight anosognosia as a barrier to rehabilitation, a risk to safe discharge, and a predictor of poorer psychological and functional outcomes for both patients and their carers. Currently, there exists a vast number of assessment methods for anosognosia after stroke, which vary from performance- and observation-based tasks to self-report and discrepancy-based interviews; clinicians working in stroke make arbitrary choices as to which of these methods to use on a case-by-case basis, risking missed cases and subsequently noncomprehensive care. This research aims to develop a new screening tool for anosognosia that can be routinely implemented with post-stroke patients in hospital settings, to inform care, rehabilitation, and discharge. The study will explore the acceptability and feasibility of the new screening tool among multi-disciplinary staff working on a stroke rehabilitation unit, and provide grounds for future studies to assess the screen's psychometric properties and ability to inform novel interventions for anosognosia. Findings will have great implications for stroke survivors, their carers, and healthcare professionals alike.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or above who are admitted to the stroke rehabilitation unit with a clinical diagnosis of stroke.
* Multi-disciplinary staff working on the stroke rehabilitation unit.

Exclusion Criteria:

* Patients with a clinical diagnosis other than stroke.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients admitted to a stroke rehabilitation ward.
  Multi-disciplinary staff working with stroke patients on a stroke rehabilitation ward.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Acceptability and Feasibility of new screening tool among multi-disciplinary staff | From recruitment, throughout 4-6 months of screen implementation, to the completion of focus groups approximately 8 months after recruitment.
  Focus groups will be conducted with staff who administer the new screening tool on the target stroke rehabilitation ward, to explore their views of and experiences with the tool. This will be in relation to the tool's content, structure, length, response/scoring formats, and administration demands.

SECONDARY OUTCOMES:
Uptake and Validity of new screening tool, with patients | Over 4-6 months, from recruitment until the completion of screen implementation.
  Demographic data and stroke-related data (stroke location, severity) will provide descriptive insight into the usability of the tool across subgroups of the sample. Numbers of completed forms will provide descriptive insight into the uptake of the screening tool. Inter-rater reliability will provide insight into the tool's equivalence.

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Clarke, DClinPsy, QiCN, Study Director — University of Exeter